CLINICAL TRIAL: NCT00878137
Title: INR Determined by Plasma-based Methods Versus Newer Point-of-care Instruments in Patients With Antiphospholipid-antibody Syndrome Treated With Anticoagulants
Brief Title: Reliability of Point-of-care INR Measurements in Patients With Antiphospholipid-antibody Syndrome Treated With Warfarin
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: International Technidyne Corporation (Industry)
Responsible Party: Principal Investigator, Lauren McKnight, PharmD, CPP, Clinical Pharmacist, University of North Carolina, Chapel Hill
Other Study IDs: POC Comparison 08-1883
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- APLA: Patients with antiphospholipid antibody syndrome.
  Interventions: Device: INR by point-of-care instruments and venopuncture
- Control: Patients on warfarin therapy but without antiphosphilipid antibody syndrome.
  Interventions: Device: INR by point-of-care instruments and venopuncture

INTERVENTIONS:
Device: INR by point-of-care instruments and venopuncture — Three fingersticks will be performed and from each one drop of capillary or venous whole blood collected from a fingerstick performed by the primary investigator to measure PT/INR using the CoaguChekXSTM (10 microliters), ProTimeTM (27 microliters), the investigational ProTime, and INRatioTM 15 microliters) point-of-care instruments and one i.v. blood draw (20 mL of blood) will be performed by a phlebotomist.

SUMMARY:
The antiphospholipid-antibody syndrome (APLA), which includes lupus anticoagulant, anticardiolipin, and anti-beta-2-glycoproteinI antibodies, is a thrombophilic disorder associated with arterial thrombosis, venous thrombosis or both. Patients diagnosed with APLA have a higher risk of recurrent thrombosis than do patients without known antibodies. Currently, warfarin is considered the anticoagulant of choice for prophylactic antithrombotic treatment for APLA patients after their first episode of thrombosis. In some patients with APLA who are treated with warfarin, the INR values determined on plasma are unreliable due to an influence of the APLA on the INR. In these individuals, alternative monitoring methods, such as factor II activity, chromogenic factor X activity or prothrombin-proconvertin time should be used to assess adequate anticoagulation. These tests are expensive and not widely available to some clinicians. Point-of-care (POC) instruments, on the other hand, are readily accessible to clinicians. Previous research has shown that INR values from 3 older point-of-care (POC) instruments are unreliable in 1/3 of APLA patients (CoaguChekTM, ProTimeTM, INRatioTM). However, there are now newer versions of these POC instruments available (CoaguChek XSTM, an investigational ProTime device, and a newer INRatioTM device) and it is unknown if these newer POC instruments are reliable in patients with APLA. The purpose of this study is to determine whether newer POC instruments are reliable in patients with APLA.

ELIGIBILITY:
APLA Inclusion Criteria:

* Prolongation of a phospholipid-dependent screening assay, 2) lack of correction of a prolonged screening assay after a 1:1 mix with pooled normal plasma, and 3) correction of a prolonged screening assay by the addition of excess phospholipid. Two positive lupus anticoagulant confirmations at least 3 months apart will be required.
* Diagnosis of anticardiolipin antibodies defined as elevated levels of ACA-IgG (>30) and/or ACA-IgM (>15) on two separate occasions at least 3 months apart.
* Stable warfarin therapy, defined as the maintenance of a warfarin dose for a minimal of 2 weeks regardless of INR.

APLA Exclusion Criteria:

* Patients whose warfarin dose has changed within the past 2 weeks.

Control Inclusion Criteria:

* No evidence of either a positive LA or ACA diagnosis by confirmation of negative laboratory values and/or documentation of no clinical signs and symptoms concurrent with these conditions.
* Stable warfarin therapy, defined as the maintenance of a warfarin dose for a minimal of 2 weeks regardless of INR.

Control Exclusion Criteria:

* Patients whose warfarin dose has changed within the past 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: APLA patients will be identified through the UNC Thrombophilia Program database. Control patients will be recruited at UNC Anticoagulation Clinic visits.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B McKnight, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States